CLINICAL TRIAL: NCT01718587
Title: Difference in Efficacy Between Umbilical Cord Mesenchyma Stem Cell Transplantation and Classical Therapy in Liver Cirrhosis Patients
Brief Title: Difference in Efficacy Between Stem Cell Transplantation and Classical Therapy in Liver Cirrhosis Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Collaborators: The First Hospital of Hebei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-10-09 TC liver cirrhosis
Record Dates: First submitted 2012-10-25; First posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Liver Cirrhosis
Keywords: umbilical cord mesenchyma stem cell; liver cirrhosis; antiviral therapy
MeSH Terms: conditions — Liver Cirrhosis | interventions — Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stem cell transplantation therapy (Experimental): umbilical cord mesenchyma stem cell transplantation through interventional procedures do in liver cirrhosis patients.
  Interventions: Procedure: stem cell transplantation through interventional procedure
- antiviral therapy (Active Comparator): Antiviral therapy: lamivudine, 100 mg per day (oral dose); or adefovir dipivoxil 10 mg per day (oral dose); or grace entecavir 0.5-1mg per day (oral dose); or behalftelbivudine 600 mg per day (oral dose).
  Supportive therapy are allowed to use on patients not including intravenous infusions of plasma or albumin.
  Interventions: Drug: antiviral therapy (lamivudine, other antiviral drugs)

INTERVENTIONS:
Procedure: stem cell transplantation through interventional procedure — interventional procedure once
  Other Names: UCMSC transplantation
  Arms: stem cell transplantation therapy
Drug: antiviral therapy (lamivudine, other antiviral drugs) — lamivudine, 100 mg per day (oral dose); or adefovir dipivoxil 10 mg per day (oral dose); or grace entecavir 0.5-1mg per day (oral dose); or behalftelbivudine 600 mg per day (oral dose).
  Other Names: lamivudine or other antiviral drugs.
  Arms: antiviral therapy

SUMMARY:
The current treatment methods of liver cirrhosis are limited ,including antiviral therapy,supportive therapy and liver transplantation. Antiviral therapy and Supportive therapy especially the regularly intravenous infusions of plasma or albumin are combined in the clinical classical therapy treatment. In the other hand,umbilical cord mesenchyma stem cell with self and directed differentiation capacity can effectively rescue experimental liver failure and contribute to liver regeneration, which suggests the feasibility of stem cell transplantation therapy. In this study, the safety and efficacy of umbilical cord mesenchyma stem cell transplantation through interventional procedures and classical therapy in patients liver cirrhosis will be evaluated and compared.

DETAILED DESCRIPTION:
This study will includ two research centers, the number of patients in transplantation group will be 30, the number of patients in classical therapy group will be 30. All the inclusion and exclusion criteria will be same and the data analysis will be complete by the epidemiological commissioner.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of liver cirrhosis;
* Without hepatic encephalopathy;
* No ascites or have easily dissipated ascites;
* Value of bilirubin is less than 100;
* Value of albumin is greater than 16 g / L;
* Prothrombin time is less than 21 seconds;

Exclusion Criteria:

* Severe cardiovascular disease, and immunocompromised patients;
* Patients with localized lesions affecting graft infection;
* Coagulation disorders;
* Liver nodules more than 2cm or Liver cancer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-05 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
liver volume calculated by MRI | baseline
  Instrument:universal 1.5 Tesla superconducting MRI instrument. Slice thickness :2mm.
change from baseline in liver volume calculated by MRI at 6 months | 6 months after treatment
  Instrument:universal 1.5 Tesla superconducting MRI instrument. Slice thickness :2mm.
change from baseline in liver volume calculated by MRI at 12 months | 12 months after treatment
  Instrument:universal 1.5 Tesla superconducting MRI instrument. Slice thickness :2mm.

SECONDARY OUTCOMES:
blood biochemistry | baseline, 1,3,6 and 12 months after treatment or transplantation
  1. alanine aminotransferase
  2. aspartate aminotransferase
  3. gamma-glutamyltransferase(GGT)
  4. alkaline phosphatase
  5. total bilirubin
  6. direct bilirubin
  7. The total bile acid (TBA)
  8. albumin
  9. the proportion of white balls
blood test | baseline,1,3,6 and 12 months after treatment or transplantation
  1. platelet count (PLT)
  2. mean platelet volume (MPV)
  3. platelet distribution width (PDW)
  4. platelet hematocrit (PCT)
  5. alpha feto protein (AFP)
liver enzyme fiber spectrum | baseline,1,3,6 and 12 months after treatment or transplantation
  1. laminin (LN)
  2. Ⅳ collagen detection (CIV)
  3. hyaluronic acid (HA)
  4. procollagen Ⅲ(PC Ⅲ)
coagulation | baselin,1,3,6 and 12 months after treatment or transplantation
  1. prothrombin time (PT)
  2. activated partial thromboplastin time (APTT)
  3. fibrinogen (FIB)
  4. thrombin time (TT)
portal vein and splenic vein measure | baseline,1,3,6 and 12 months after treatment or transplantation
  1)Portal vein diameter (Dpv) 2）Portal vein maximum velocity (Vmaxpv) 3）Portal vein blood flow per minute (Qpv) 4) The splenic vein diameter (Dsv) 5) Splenic vein maximum flow velocity (Vmaxsv) 6) Splenic vein blood flow per minute (Qsv)
estrogen and progestin in blood | baseline,1,3,6 and 12 months after treatment or transplantation
  estrogen and progestin

OTHER OUTCOMES:
liver biopsy | baseline,6 and 12 months after transplantation
  The result of liver biopsy judged by the same one expert.
gastroscopy | baseline,6 and 12 months after treatment or transplantation
  Observe and photograph the related varicose veins.

CONTACTS AND LOCATIONS:
Overall Officials: Yihua An, PhD, Study Director — Department of Stem Cell Transplantation, the General Hospital of Chinese People's Armed Police Force
Locations (1):
- Yihua An, Beijing, China